CLINICAL TRIAL: NCT07203989
Title: The Effect of Video Calls With Family Members During Operating Room Waiting on Stress, Anxiety, and Surgical Fear in Patients Undergoing Transurethral Resection of Bladder Tumor: A Multicenter Randomized Controlled Trial
Brief Title: The Effect of Video Calls With Family Members During Operating Room Waiting on Stress, Anxiety, and Surgical Fear in Patients Undergoing Transurethral Resection of Bladder Tumor
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Erdogan Yakit, Lecturer, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HKU-2025-TURBT-FV-RCT01
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Bladder Tumor (TURBT); Bladder (Urothelial, Transitional Cell) Cancer
Keywords: Transurethral resection of bladder tumor (TURBT); Preoperative anxiety; Surgical fear; Family-centered care; Video call intervention
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - Intervention Group (Experimental): Family Meeting:Patients will have a real-time video call with one designated family member while waiting in the operating room before anesthesia induction. The call will last until anesthesia preparation begins.
  Interventions: Behavioral: family-supported care
- Control Group (No Intervention): Standard Maintenance: Patients will undergo the standard surgical preparation and waiting process in the operating room without any contact with family members.

INTERVENTIONS:
Behavioral: family-supported care — Family video calling in the operating room
  Other Names: Family video calling in the operating room
  Arms: Experimental - Intervention Group

SUMMARY:
This study aims to investigate the effect of video calls with family members during the preoperative waiting period in the operating room on stress, anxiety, and surgical fear in patients undergoing transurethral resection of bladder tumor (TURBT). Bladder cancer is a common urological malignancy, and psychological problems are frequently observed in the preoperative period. The absence of family support in the operating room may increase anxiety and fear, triggering physiological stress responses and raising the risk of complications.

This multicenter randomized controlled trial will be conducted between September 2025 and March 2027 at Bitlis State Hospital and Tatvan State Hospital. The study sample will include 128 eligible patients, randomly assigned to intervention and control groups. Patients in the intervention group will have a video call with a designated family member in the operating room, while control group patients will receive routine care.

Data will be collected using the Descriptive Information Form, the Surgical Fear Questionnaire, and the Visual Analogue Scale; stress levels will be assessed through serum cortisol and glucose values. Measurements will be taken at three time points: preoperatively (T0), immediately before anesthesia (T1), and on the first postoperative day (T2).

The study is expected to demonstrate that maintaining family support through video calls in the preoperative period reduces anxiety, fear, and stress, thereby improving surgical outcomes and contributing to the development of family-centered care practices.

DETAILED DESCRIPTION:
This study investigates the effect of family-supported video calls on patients with bladder tumor scheduled for transurethral resection (TURBT) during the preoperative waiting period in the operating room. Preoperative anxiety, surgical fear, and stress are common among surgical patients and may negatively influence physiological responses and postoperative outcomes. Allowing real-time communication with a family member through a secure digital platform may provide psychological support, reduce anxiety and fear, and mitigate stress-related physiological changes.

The study is designed as a multicenter randomized controlled trial conducted at Bitlis State Hospital and Tatvan State Hospital between September 2025 and March 2027. Eligible patients will be randomly assigned to either the intervention group, who will have a structured video call with a designated family member before anesthesia induction, or the control group, who will receive standard preoperative care without family contact in the operating room. Outcomes will include anxiety, surgical fear, and stress levels, measured using validated scales and physiological parameters. Findings from this study are expected to contribute to the development of family-centered care strategies aimed at improving perioperative psychological well-being and surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to read and write in Turkish
* Scheduled for transurethral resection of bladder tumor (TURBT)
* Has a family member, friend, or relative able to participate in video calls
* The accompanying family member or relative has a device suitable for video calls (smartphone, tablet, etc.)
* Has waited at least 20 minutes in the operating room before surgery
* No hearing, speech, or language-related communication barriers
* No psychological disorders that could affect fear or anxiety
* Not using medications that could alter fear or anxiety levels
* Scheduled for surgery between 08:00 and 12:00
* Willing to voluntarily participate in the study

Exclusion Criteria:

* Surgery is canceled after the patient has been enrolled in the study
* Patient chooses to withdraw from the study after enrollment
* Individuals with any diagnosed chronic disease
* Experiencing connection problems during the video call
* Patients who receive premedication during the waiting period to relieve anxiety

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety Level (Visual Analogue Scale) | Anxiety levels will be measured at three different time points: T0: On the morning of the surgery, at 08:00 in the ward T1: In the operating room, immediately before anesthesia induction T2: The morning after the surgery, at 08:00
  Anxiety levels will be assessed using the Visual Analogue Scale (VAS), scored from 0 (no anxiety) to 10 (worst possible anxiety). Higher scores indicate greater anxiety.
stress | Blood samples will be collected from patients at three different times. • T0: On the morning of surgery, in the ward at 8:00 a.m. • T1: In the operating room, just before anesthesia induction • T2: The day after surgery, at 8:00 a.m.
  Serum cortisol and serum glucose levels will be measured to determine patients' stress levels. Increases in cortisol and glucose levels indicate increased stress levels.
Surgical Fear Level | Patients' surgical fear levels will be measured at two different times. • T0: On the morning of surgery, in the ward at 8:00 a.m. • T1: In the operating room, just before anesthesia induction
  The Surgical Fear Scale (SFS) will be used to determine the level of fear in patients.
  Surgical Fear Scale: The Surgical Fear Scale was first developed by Theunissen et al. in 2014 to determine the level of surgical fear in patients undergoing surgery.
  The Surgical Fear Scale consists of eight items and two subscales, scored from 0 to 10. The first four items measure fear of short-term surgical outcomes, and the last four items measure fear of long-term outcomes. Each subscale is aggregated, and the sum of the two subscale scores constitutes the total scale score. The total score for the scale ranges from 0 to 80. Low scores indicate low levels of surgical fear, while high scores indicate high levels of surgical fear.

CONTACTS AND LOCATIONS:
Overall Officials: Erdoğan YAKIT, Study Chair — BİTLİS EREN UNİVERSTY
Locations (2):
- Turkey (Türkiye) (2):
  - Tatvan State Hospital, Bitlis, Turkey, Bitlis, Tatvan
  - Bitlis State Hospital, Bitlis, Turkey, Bitlis

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to patient confidentiality and privacy concerns, as well as institutional regulations regarding clinical data handling.